CLINICAL TRIAL: NCT04173286
Title: Is Short Antibiotherapy Duration After Drainage Suitable for Patients Admitted in Intensive Care Medicine With a Severe Acute Cholangitis?
Acronym: CASCAD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC19_0423
Record Dates: First submitted 2019-11-20; First posted 2019-11-21 (Actual); Last update posted 2019-11-21 (Actual); Status verified 2019-11

CONDITIONS: Acute Cholangitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- short term antibiotics: < 7 days
  Interventions: Procedure: antibiotherapy
- long terms antibiotics: > 7 days
  Interventions: Procedure: antibiotherapy

INTERVENTIONS:
Procedure: antibiotherapy — < 7 days

SUMMARY:
Acute cholangitis (AC) occurs when biliary stenosis, due to various benign causes (often gallstones) or the presence of a tumour, leads to cholestasis and biliary infection. AC is a life-threatening infection if not diagnosed and treated in time, its mortality ranges from 1.4% to 5.2%. AC can be classified into different stages of severity depending on organ failure. A severity classification has been proposed by the Asian recommendations of Tokyo 2013: Grade I (Benin), Grade II (Moderate) and Grade III (Severe).

AC treatment includes endoscopic or percutaneous bile drainage in combination with systemic antibiotic treatment. It is currently recommended that patients with severe CA (Grade III) have biliary drainage within 24 hours, although it has not been shown to improve their survival. The emergence of antibiotic-resistant germs, which is a public health issue, calls for reasonable and considered use of antibiotics. Reducing the duration of antibiotic therapy is a fundamental measure of antimicrobial management and antibiotics sparing. 7 to 10 days of antibiotic treatment is common in the treatment of CA. A 14-day treatment is recommended in case of associated bacteremia. A recent study of 263 patients showed that reducing the duration of antibiotic therapy to less than 7 days in patients with CA associated with bacteremia with effective drainage does not increase the risk of recurrence or mortality at 30 days. However, this study was monocentric retrospective and compared groups that were unbalanced in terms of CA severity. The optimal duration of antibiotic therapy in the treatment of CA in critically ill patients hospitalized in intensive care remains poorly known.

The main purpose of this study is to compare short antibiotic therapy with long antibiotic therapy in terms of mortality in patients with AC admitted in intensive care unit (ICU).

DETAILED DESCRIPTION:
Using electronic patient data monitoring systems, the investigators reviewed all patients with a diagnosis of AC admitted to digestive liver disease unity or ICUs at the Nantes University Hospital, Rennes University Hospital from January 1, 2006, to december 31, 2018. For enrolled patients, general clinical characteristics were collected. Patients were categorized into two groups according to antibiotics duration, and the differences of these characteristics between two groups were evaluated.

ELIGIBILITY:
Inclusion Criteria:

Adult patients (age >18 years) with acute cholangitis Admitted in Intensive care units With a successful biliary drainage And treated with antibiotics

Exclusion Criteria:

patients under 18 years unable to receive a drainage or inefficient drainage Patients with a decision to limit care at the admission pregnancy

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Major patient, hospitalized in a MIR with a diagnosis of CA between 2006 and 2019, whatever the etiology, having had a drainage of the bile ducts regardless of the technique used and the initiation of antibiotic therapy.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2019-10-07 (Actual); Primary Completion 2020-01-01 (Estimated); Study Completion 2021-01-01 (Estimated)

PRIMARY OUTCOMES:
mortality | day 28
  Comparison of mortality at day 28 between the two group.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Nantes, Nantes, France